CLINICAL TRIAL: NCT02017379
Title: Randomized Control Trial Comparing Prokinetics and Their Influence on Endoscopy Outcomes for Upper GI Bleed.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not recruit any subjects
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: E13018
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: upper gastrointestinal bleeding; melena; hematemesis
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Melena; Hematemesis | interventions — Erythromycin; Erythromycin Estolate; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (3):
- Erythromycin (Experimental): Intravenous erythromycin infusion (dose: 250 mg) 30 min-60 min before procedure
  Interventions: Drug: Erythromycin
- Metoclopromide (Experimental): Intravenous metoclopromide infusion (dose: 10 mg) 30-60 minutes prior to endoscopy
  Interventions: Drug: Metoclopromide
- Control (No Intervention): no medications will be given prior to endoscopy

INTERVENTIONS:
Drug: Erythromycin
  Other Names: Erythrocin, E-Mycin, Ery-Tab, Ilosone
  Arms: Erythromycin
Drug: Metoclopromide
  Other Names: Reglan, Maxolon, Metozolv ODT
  Arms: Metoclopromide

SUMMARY:
This is a study comparing the effect of erythromycin or metoclopramide, 2 prokinetic drugs (Drugs which are known to speed up the emptying of the stomach or in other words to move the blood out of the stomach faster) given before endoscopy to patients with upper Gastrointestinal bleeding compared to patients who will not receive either of these medications before their endoscopy.

DETAILED DESCRIPTION:
To compare the efficacy of pre-endoscopic interventions namely erythromycin, metoclopromide vs control in improving the outcomes of endoscopy in ICU patients admitted upper GI bleeding.

Specific aims:

1. Wither erythromycin, metoclopromide vs control can enable visualization of the entire gastric mucosa .
2. Wither erythromycin, metoclopromide vs control can improve the quality of stomach and duodenum visualization: using the scoring system by Fossard et al

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-80)
* who are admitted to the ICU for hematemesis, or coffee ground emesis

Exclusion Criteria:

1. Patients younger than 18 yrs old or older than 80 yrs
2. Patients who refuse to consent to be in our study
3. Pregnant patients
4. Prior use of prokinetics in the last 48 hours
5. History of cardiac arrhythmia
6. Allergy to erythromycin or metoclopromide
7. Patients with QT prolongation (query 7)

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed O Othman, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Science Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Erythromycin: Intravenous erythromycin infusion (dose: 250 mg) 30 min-60 min before procedure
  Erythromycin
- Metoclopromide: Intravenous metoclopromide infusion (dose: 10 mg) 30-60 minutes prior to endoscopy
  Metoclopromide
Period: Overall Study
Arm/Group | Erythromycin | Metoclopromide | Control
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythromycin | Metoclopromide | Control | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Erythromycin, Metoclopromide vs Control Enabling Visualization of the Entire Gastric Mucosa .
Description: Whether erythromycin, metoclopramide versus control can enable visualization of the entire gastric mucosa .
Time Frame: 45 minutes
Population: as for baseline characteristics
Arm/Group | Erythromycin | Metoclopromide | Control
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Erythromycin, Metoclopromide vs Control Improving the Quality of Stomach and Duodenum Visualization
Description: Whether erythromycin, metoclopramide vs control can improve the quality of stomach and duodenum visualization: using the scoring system by Fossard et al
Time Frame: 45 minutes
Population: as for baseline characteristics
Arm/Group | Erythromycin | Metoclopromide | Control
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Source of Bleeding
Description: Ability to identify the source of bleeding
Time Frame: 45 minutes
Population: as for baseline characteristics
Arm/Group | Erythromycin | Metoclopromide | Control
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Second-look Endoscopy
Description: Need for second-look endoscopy
Time Frame: 48 hours
Population: as for baseline characteristics
Arm/Group | Erythromycin | Metoclopromide | Control
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Blood Units Transfused
Description: Mean number of blood units transfused
Time Frame: 48 hours
Population: as for baseline characteristics
Arm/Group | Erythromycin | Metoclopromide | Control
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Mortality
Description: All cause mortality
Time Frame: 30 days
Population: as for baseline characteristics
Arm/Group | Erythromycin | Metoclopromide | Control
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Description: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | Erythromycin | Metoclopromide | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes